CLINICAL TRIAL: NCT01717833
Title: The Role of Neuromuscular Electrical Stimulation as a Tool for Post ICU Rehabilitation
Brief Title: The Role of NEMS for Post ICU Rehabilitation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Serafim Nanas, Professor, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SN01032010
Record Dates: First submitted 2012-10-21; First posted 2012-10-31 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Critical Illness
Keywords: ICU acquired weakness; Critical illness polyneuromyopathy; post ICU rehabilitation; neuromuscular electrical rehabilitation; handgrip
MeSH Terms: conditions — Critical Illness | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NEMS group (Experimental)
  Interventions: Procedure: NEMS
- Sham group (Sham Comparator)
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: NEMS — NEMS sessions on both lower extremities (quadriceps and peroneus longus) simultaneously
  Other Names: Neuromuscular Electrical stimulation
  Arms: NEMS group
Procedure: Sham — Sham sessions of neuromuscular electrical stimulation
  Other Names: Sham neuromuscular electrical stimulation
  Arms: Sham group

SUMMARY:
The purpose of this study is to investigate the role of NEMS as a rehabilitation tool for muscle weakness following critical illness. The investigators hypothesized that NEMS combined with exercise rehabilitation will have a beneficial role in restoration of muscle strength

DETAILED DESCRIPTION:
Survivors of critical illness are presented with significant physical impairment that is associated with reduced functional ability and health -related quality of life both in the short and long-term.

Neuromuscular electrical stimulation (NEMS) has been proposed as an alternative exercise modality in patients with severe chronic obstructive pulmonary disease and chronic heart failure, who cannot perform active exercise. NEMS has also been used as a preventive tool for intensive care unit (ICU) acquired weakness (ICUAW). Its role as a tool for post ICU rehabilitation has not been evaluated so far.

A randomized intervention study was designed to assess the efficacy of NEMS, as a rehabilitative tool for critical illness survivors. The first day that patients are discharged from the ICU after stratified randomization are assigned to the NEMS group or to the control group. In the NEMS group, NEMS will be applied to both lower extremities of the NEMS -group simultaneously (quadriceps femoris muscle and peroneus longus) on a daily basis, along with a personalized exercise program. NEMS sessions will continue until patient discharge from hospital. In the control group, sham NEMS will be applied along with standard care when it comes to physiotherapy. At hospital discharge patients of both groups of will receive a rehabilitation booklet. Patients on the NEMS group that have significant muscle weakness will have NEMS sessions at home for a period of 2 months. Patients are evaluated at 3 and 6 months after hospital discharge

ELIGIBILITY:
Inclusion Criteria:

* Patients under mechanical ventilation for> 72hours during ICU stay
* Patients able to perform simple commands (able to be evaluated by MRC scale)

Exclusion Criteria:

* age < 18 > 85 years
* pregnancy
* pre-existing neuromuscular disease (e.g. Gravis)
* fractures or skin lesions that do not allow the implementation of NEMS
* presence of pacemaker or defibrillator
* fractures of spine that so not allow mobilization
* BMI > 35 kg/m2
* terminal disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | up to 2.5 years

SECONDARY OUTCOMES:
Duration of hospital stay | up to 2.5 years
Functional ability | up to 2.5 years
  Functional ability will be assessed with the FIM score
Quality of life | up to 2.5 years

OTHER OUTCOMES:
Muscle strength in patients with ICU acquired weakness (ICUAW) at ICU discharge | up to 2.5 years
  In the subgroup of patients diagnosed with ICUAW improvement in muscle strength will be assessed in patients of the NEMS group as compared to the sham-NEMS group

CONTACTS AND LOCATIONS:
Overall Officials: Serafim Nanas, Professor, Principal Investigator — University of Athens
Locations (1):
- First Critical Care Unit, Evaggelismos Hospital, School of Medicine, Athens, Greece

REFERENCES:
- [Derived] Patsaki I, Gerovasili V, Sidiras G, Karatzanos E, Mitsiou G, Papadopoulos E, Christakou A, Routsi C, Kotanidou A, Nanas S. Effect of neuromuscular stimulation and individualized rehabilitation on muscle strength in Intensive Care Unit survivors: A randomized trial. J Crit Care. 2017 Aug;40:76-82. doi: 10.1016/j.jcrc.2017.03.014. Epub 2017 Mar 22. PMID 28364678